CLINICAL TRIAL: NCT05396833
Title: An Open-label, Multicenter Phase Ib Study of the Safety, Tolerability, and Pharmacokinetic/Pharmacodynamic Profile of the ATR Inhibitor Tuvusertib (M1774) in Combination With DNA Damage Response Inhibitors or Immune Checkpoint Inhibitors in Patients With Metastatic or Locally Advanced Unresectable Solid Tumors (DDRiver Solid Tumors 320)
Brief Title: Study of Tuvusertib (M1774) in Combination With DNA Damage Response Inhibitor or Immune Checkpoint Inhibitor (DDRiver Solid Tumors 320)
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: EMD Serono Research & Development Institute, Inc. (Industry)
Collaborators: Merck KGaA, Darmstadt, Germany (Industry)
Responsible Party: Sponsor
Organization: EMD Serono (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MS201924_0020; 2022-500287-35-00 (Other: EU Trial Number)
Record Dates: First submitted 2022-05-24; First posted 2022-05-31 (Actual); Last update posted 2025-09-26 (Actual); Status verified 2025-09

CONDITIONS: Metastatic or Locally Advanced Unresectable Solid Tumors
Keywords: ATR inhibitor; ATM inhibitor; Immunotherapy; Tuvusertib (M1774); Lartesertib (M4076); Avelumab; Metastatic or Locally Advanced Unresectable Solid Tumors; DNA Damage Response Inhibitor; Immune Checkpoint Inhibitor
MeSH Terms: conditions — Neoplasm Metastasis | interventions — avelumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (7):
- Part A1: Tuvusertib and Lartesertib (Experimental)
  Interventions: Drug: Tuvusertib; Drug: Lartesertib
- Part A1.1: Tuvusertib and Lartesertib (Experimental): Assessment of the Effect of Food (Low-fat Meal) on the PK of M4076 Monotherapy Followed by Treatment with M1774 in Combination with M4076
  Interventions: Drug: Tuvusertib; Drug: Lartesertib
- Part A1.2: Tuvusertib and Lartesertib (Experimental): Relative Bioavailability Assessment of Tuvusertib Tablet (TF1) vs Capsule Followed by Treatment with Tuvusertib in Combination with Lartesertib
  Interventions: Drug: Tuvusertib; Drug: Lartesertib
- Part A2: Tuvusertib and Lartesertib (Experimental): ATM in prostate cancer (Part A2)
  Interventions: Drug: Tuvusertib; Drug: Lartesertib
- Part A3: Tuvusertib and Lartesertib (Experimental): ARID1A in endometrial cancer
  Interventions: Drug: Tuvusertib; Drug: Lartesertib
- Part A2/A3: Tuvusertib and Lartesertib (Experimental): Tablet formulation (TF1, test) compared to a capsule formulation (reference)
  Interventions: Drug: Tuvusertib; Drug: Lartesertib
- Part B1: Tuvusertib and Avelumab (Experimental)
  Interventions: Drug: Tuvusertib; Drug: Avelumab

INTERVENTIONS:
Drug: Tuvusertib — Tuvusertib will be administered orally once daily over a defined period of time in Part A1, A1.1, A1.2, A2, A3, A2/A3, and Part B1 until disease progression, death, discontinuation, or end of study.
  Other Names: M1774
Drug: Lartesertib — Lartesertib will be administered orally once daily over a defined period of time in Part A1, A1.1, A1.2, A2, A3, A2/A3, until disease progression, death, discontinuation, or end of study.
  Other Names: M4076
  Arms: Part A1.1: Tuvusertib and Lartesertib; Part A1.2: Tuvusertib and Lartesertib; Part A1: Tuvusertib and Lartesertib; Part A2/A3: Tuvusertib and Lartesertib; Part A2: Tuvusertib and Lartesertib; Part A3: Tuvusertib and Lartesertib
Drug: Avelumab — Avelumab will be administered by intravenous infusion once a day over a defined period of time in Part B1 until disease progression, death, discontinuation, or end of study.
  Arms: Part B1: Tuvusertib and Avelumab

SUMMARY:
This is an open-label, multicenter, clinical study conducted in multiple parts to establish the safety, tolerability, Pharmacokinetic/Pharmacodynamic (PK/PD) profile, maximum tolerated dose (MTD) combinations (if observed) and recommended dose for expansion (RDE) combination for tuvusertib in combination with lartesertib (in Part A1), food effect on the PK of lartesertib as monotherapy followed by treatment with tuvusertib in combination with lartesertib in participants with specific tumor types (in Part A1.1), relative bioavailability of a tuvusertib tablet formulation vs capsule formulation followed by treatment with tuvusertib (capsule) in combination with lartesertib in participants with specific tumor types (in Part A1.2), safety/tolerability and early signs of clinical activity of tuvusertib (capsule)and lartesertib in combination in participants with prostate cancer harboring loss of function (LoS) mutation in the gene ATM based on historic data collected prior to prescreening in circulating tumor (ct) DNA (liquid biopsies) or tumor biopsies (in Part A2), safety/tolerability and early signs of clinical activity of tuvusertib and lartesertib in combination in participants with endometrial cancer harboring LoS mutation(s) in the gene ARID1A based on historic data collected prior to prescreening in ctDNA (liquid biopsies) or tumor biopsies (in Part A3), the relative bioavailability of a tuvusertib tablet formulation (TF1, test) compared to a capsule formulation (reference) will also be investigated (in Part A2/A3), and identify a potential set of MTD combinations, and establish the RDE for the combination of tuvusertib and avelumab in participants with metastatic or locally advanced unresectable solid tumors (in Part B1).

ELIGIBILITY:
Inclusion Criteria:

* Parts A1, A1.1, A1.2, A2, A3, and A2/3: Participants with metastatic or locally advanced unresectable solid tumors refractory to standard therapy or for which no standard therapy is judged appropriate by the Investigator, which may convey clinical benefit, or who cannot tolerate standard of care treatment
* Parts A1.1 and A1.2: Triple negative breast cancer, epithelial ovarian cancer, castrate resistant prostate cancer, urothelial cancer, endometrial cancer, and colorectal cancer independent of mutation status.
* Part A2: Participants with advanced prostate cancer whose tumor carries a genetic loss of function (LoF) mutation(s) in the gene ataxia telangiectasia mutated (ATM). No more than 3 prior lines of therapy for castrate resistant disease. Prior therapy must have included a taxane and a novel antiandrogen (example [e.g.] enzalutamide).
* Part A3: Participants with advanced endometrial cancer whose tumor carries a genetic LoF mutation(s) in the gene AT-rich interaction domain 1A (ARID1A). Prior therapy must have included a platinum agent. Prior therapy must also have included a checkpoint inhibitor if the participant has mismatch repair (MMR)-deficient endometrial cancer. Note for Parts A2/A3: Participants with ATM LoF mutated prostate cancer and ARID1A LoF mutated endometrial cancer should be prioritized to the respective expansion arms instead of being enrolled in Part A1.1. The presence of ATM and ARID1A LoF mutations will be determined according to historic data collected prior to prescreening, generated by an assay with appropriate regulatory status, in either tumor or liquid biopsy. The Sponsor will confirm that mutations certified by historic data fulfil this definition.
* Participants with eastern Cooperative Oncology Group (ECOG) performance status 0 or 1, with estimated life expectancy of at least 3 months
* Adequate hematological, hepatic, and renal function as defined in the protocol
* Other protocol defined inclusion criteria could apply

Exclusion Criteria:

* Participants with any condition, including any uncontrolled disease state other than with metastatic or locally advanced unresectable solid tumors, that in the Investigator's opinion constitutes an inappropriate risk or a contraindication for participation in the study or that could interfere with the study objectives, conduct, or evaluation
* Participants with a known additional malignancy that is progressing and/or requires active treatment
* Participants with carcinomatous meningitis are excluded regardless of clinical stability
* Participants with serious gastrointestinal bleeding within 3 months, refractory nausea and vomiting, uncontrolled diarrhea, known malabsorption, significant small bowel resection or gastric bypass surgery, use of feeding tubes, other chronic gastrointestinal disease, and/or other situations that may preclude adequate absorption of oral medications
* Participants with organ transplantation, including allogeneic stem cell transplant
* Other protocol defined exclusion criteria could apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2022-06-07 (Actual); Primary Completion 2026-04-03 (Estimated); Study Completion 2026-04-03 (Estimated)

PRIMARY OUTCOMES:
Part A1: Number of Participants With Dose-Limiting Toxicities (DLTs) During the DLT Evaluation Period | Day 1 up to Day 28
Part A1: Number of Participants With Adverse Events (AEs) and Treatment-Related AEs | Baseline up to 18 months
Part B1: Number of Participants with Dose-Limiting Toxicities (DLTs) During the DLT Evaluation Period | Day 1 up to Day 28
Part B1: Number of Participants with AEs and Treatment-Related AEs | Baseline up to 18 months
Part A1: Change From Baseline in Pharmacodynamic (PD) Biomarker | Pre-dose up to approximately 1 month
  The PD biomarker of histone variant will be measured by flow cytometry.
Part B1: Change From Baseline in PD Biomarker | Pre-dose up to approximately 1 month
  The PD biomarker of histone variant will be measured by flow cytometry.
Part A1.1: PK Plasma Concentration of Lartesertib Under Fed and Fasted Conditions | Day -1 up to Period 1 Day 1
Part A2/A3: Objective Response according to Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 as assessed by Investigator | Up to 18 months after first dose administration
Part A2/A3: Number of Participants With AEs and Treatment-Related AEs | Baseline up to 18 months
Part A1.2: Relative Bioavailability Based on Area Under the Plasma Concentration Curve From Time Zero Extrapolated to Infinity [Frel(AUC0-inf)] of Tuvusertib Test Treatment Compared to Tuvusertib Reference Treatment | Day -4 up to Period 1 Day 1
Part A1.2: Relative Bioavailability Based on Area Under the Plasma Concentration Curve From Time Zero to Last Quantifiable Concentration [Frel(AUC0-t)] of Tuvusertib Test Treatment Compared to Tuvusertib Reference Treatment | Day -4 up to Period 1 Day 1
Part A1.2: Ratio Maximum Observed Plasma Concentration (Ratio[Cmax]) of Tuvusertib Test Treatment Compared to Tuvusertib Reference Treatment | Day -4 up to Period 1 Day 1
Part A2/A3: Relative Bioavailability Based on Area Under the Plasma Concentration Curve From Time Zero Extrapolated to Infinity [Frel(AUC0-inf)] of Tuvusertib Test Treatment Compared to Tuvusertib Reference Treatment | Day -4 up to Period 1 Day 1
Part A2/A3: Relative Bioavailability Based on Area Under the Plasma Concentration Curve From Time Zero to Last Quantifiable Concentration [Frel(AUC0-t)] of Tuvusertib Test Treatment Compared to Tuvusertib Reference Treatment | Day -4 up to Period 1 Day 1
Part A2/A3: Ratio Maximum Observed Plasma Concentration (Ratio[Cmax]) of Tuvusertib Test Treatment Compared to Tuvusertib Reference Treatment | Day -4 up to Period 1 Day 1

SECONDARY OUTCOMES:
Part A1: Pharmacokinetic (PK) Plasma Concentration of Tuvusertib and Lartesertib | Pre-dose up to approximately 6 months
Parts A1.2 and B1: Pharmacokinetic (PK) Plasma Concentration of Tuvusertib | Pre-dose up to approximately 6 months
Part B1: Pharmacokinetic (PK) Serum Concentration of Avelumab | Pre-dose up to approximately 18 months
Part A1 and B1: Number of Participants with Clinically Significant Abnormalities in Digital Electrocardiogram (ECG) Measures | Baseline up to 18 months
Part A1 and B1: Objective Response (OR) According to Response Evaluation Criteria in Solid Tumor (RECIST) v1.1 | Up to 18 months after first dose administration
Part B1: Number of Participants with Any Positive Anti-Drug Antibody (ADA) of Avelumab | Baseline up to 18 months
Parts A1.1, A1.2 and A2/3: Number of Participants With AEs and Treatment-Related AEs | Baseline up to 18 months
Part A1.1: PK Plasma and Urine Concentration of Lartesertib Under Fed and Fasted Conditions | Day -1 up to Period 1 Day 1
Part A2/A3: Time to Reach Maximum Plasma Concentration (tmax) of Tuvusertib | Day -4 up to Period 1 Day 1
Part A2/A3: Duration of Response according to RECIST v1.1 | Up to 18 months after first dose administration
Part A2/A3: Clinical benefit (either OR or stable disease for 6 months or more) according to RECIST v1.1. | Up to 18 months after first dose administration
Part A2/A3: Progression Free Survival according to RECIST v1.1 modified according to the Prostate Cancer Working Group 3 (PCWG-3), assessed by Investigator | Up to 18 months after first dose administration

CONTACTS AND LOCATIONS:
Overall Officials: Medical Responsible, Study Director — Merck Healthcare KGaA, Darmstadt, Germany, an affiliate of Merck KGaA, Darmstadt, Germany
Locations (22):
- United States (8):
  - Providence Medical Foundation, Santa Rosa, California
  - University of Miami School of Medicine, Miami, Florida
  - Augusta University - formerly Georgia Regents University, Augusta, Georgia
  - The University of Kansas Medical Center Research Institute, Inc., Kansas City, Kansas
  - Carolina Urologic Research Center, Myrtle Beach, South Carolina
  - Mary Crowley Cancer Research Centers, Dallas, Texas
  - University of Texas M. D. Anderson Cancer Center - Partner, Houston, Texas
  - NEXT Oncology, San Antonio, Texas
- Australia (2):
  - Royal North Shore Hospital, St Leonards
  - Calvary Mater Newcastle - PARENT, Waratah
- Princess Margaret Cancer Centre, Toronto, Canada
- South Korea (6):
  - Seoul National University Bundang Hospital, Seongnam-si
  - Severance Hospital, Yonsei University Health System - Division of Infectious Diseases, Seoul
  - Asan Medical Center, Seoul
  - Samsung Medical Center, Seoul
  - The Catholic University of Korea, Seoul St. Mary's Hospital, Seoul
  - Korea University Guro Hospital, Seoul
- Spain (5):
  - Hospital QuironSalud Barcelona - Next Oncology, Barcelona
  - Hospital Clinic de Barcelona - Servicio de Oncologia, Barcelona
  - Centro Integral Oncologico Clara Campal - Unidad de Fase I-Oncologica, Madrid
  - Hospital Universitario Quironsalud Madrid - NEXT Oncology, Madrid
  - Hospital Universitario Fundacion Jimenez Diaz - START Madrid FJD - Oncology Phase I, Madrid

IPD SHARING:
Plan to Share IPD: No
We are committed to enhancing public health through responsible sharing of clinical trial data. Following approval of a new product or a new indication for an approved product in both the US and the European Union, the study sponsor and/or its affiliated companies will share study protocols, anonymized patient data and study level data, and redacted clinical study reports with qualified scientific and medical researchers, upon request, as necessary for conducting legitimate research. Further information on how to request data can be found on our website bit.ly/IPD21

REFERENCES:
- See also: Trial Awareness and Transparency website — https://clinicaltrials.emdgroup.com/en/trial-details/?id=MS201924_0020
- See also: US Medical Information website, Medical Resources — https://medical.emdserono.com/en_US/home.html